CLINICAL TRIAL: NCT07165210
Title: A Prospective Observational Study of Left Tracheobronchial Lymph Node Metastasis in Patients With Esophageal Cancer
Brief Title: Incidence of 106TBL Lymph Node Metastasis
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director, Institute of Thoracic Oncology, Fudan University, Fudan University
Other Study IDs: ECTOP-2010
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Cancer
Keywords: lymph node metastasis; esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- prospective observation cohort: All patients who had surgery due to esophageal cancer with curative intent, no intervention was applied.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — no intervention was applied in this cohort

SUMMARY:
the study was to document the incidence of left tracheobronchial lymph node metastasis, and the risk factors of metastasis.

DETAILED DESCRIPTION:
Although the survival of esophageal cancer patients has improved with the application of chemotherapy, radiotherapy, and immunotherapy, esophageal surgery remains one of the procedures with a high risk of postoperative complications, despite significant advancements in surgical techniques in recent years.

curative surgery includes tumor resection, digestive tract reconstruction, and thorough lymph node dissection. Our previous studies demonstrated that complete right thoracic lymph node dissection significantly improves long-term survival compared to incomplete left thoracic dissection (1). However, extended three-field lymph node dissection did not show survival benefits over conventional two-field dissection (2). Therefore, the precise scope of two-field lymph node dissection in esophageal cancer requires further refinement.

Current preoperative diagnostic methods for lymph node metastasis in esophageal cancer suffer from limited sensitivity (3). In traditional two-field dissection, removing the left tracheobronchial lymph nodes may compromise blood supply to the trachea and bronchi, increase the risk of recurrent laryngeal nerve injury, and elevate postoperative complications such as cough and pneumonia. Our retrospective study on left tracheobronchial lymph node (106TBL) metastasis revealed a low transfer rate of approximately 2% (4). The risk factors for 106TBL metastasis and its long-term prognostic impact remain unclear, necessitating prospective studies to validate the necessity of this nodal station dissection.

This study aims to prospectively investigate the incidence and risk factors of tracheobronchial lymph node metastasis within the conventional dissection range, providing robust evidence for personalized treatment strategies in esophageal cancer.

Reference:

1. Li B, Hu H, Zhang Y, et al. Extended Right Thoracic Approach Compared With Limited Left Thoracic Approach for Patients With Middle and Lower Esophageal Squamous Cell Carcinoma: Three-year Survival of a Prospective, Randomized, Open-label Trial. Ann Surg . 2018 May;267(5):826-832.
2. Li B, Zhang Y, Miao L, et al. Esophagectomy With Three-Field Versus Two-Field Lymphadenectomy for Middle and Lower Thoracic Esophageal Cancer: Long-Term Outcomes of a Randomized Clinical Trial. J Thorac Oncol . 2021 Feb;16(2):310-317.
3. Li B, Li N, Liu S, et al. Does [18F] fluorodeoxyglucose-positron emission tomography/computed tomography have a role in cervical nodal staging for esophageal squamous cell carcinoma? J Thorac Cardiovasc Surg . 2020 Aug;160(2):544-550.
4. Lin K, Li B, Sun Y, et al. Precise pattern of lymphatic spread of esophageal squamous cell carcinoma: results of 1074 patients with N1 disease. J Cancer Res Clin Oncol . 2023 Nov;149(17):15819-15825

ELIGIBILITY:
Inclusion Criteria:

* patients with esophageal squamous cell carcinoma
* clinical staging: cT1-4a N0/+ M0.
* no history of other malignancy.

Exclusion Criteria:

* esophageal cancer in the neck
* poor physical status to have esophagectomy.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: observation study population
Sampling Method: Probability Sample
Enrollment: 1852 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2027-07-21 (Estimated); Study Completion 2030-07-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of left tracheobronchial lymph node metastasis | 2 years
  number of patients who had left tracheobronchial lymph node metastasis/number of patients who had resection of left tracheobronchial lymph node

SECONDARY OUTCOMES:
Risk factors of left tracheobronchial lymph node metastasis | 2 years
  risk factors that related to the metastasis of left tracheobronchial lymph node.
Survival of patients with left tracheobronchial lymph node metastasis | 5 years
  the disease-free survival and overall survival of patients who had left tracheobronchial lymph node metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
incidence, risk factors and survival data could be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the IPD and supporting information will be available from January 1st 2027 to December 31st 2030.